CLINICAL TRIAL: NCT07169877
Title: Does a Minimally Invasive Approach to Liver Resection Improve Postoperative Outcomes?
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Michael Leitman, Dean for Graduate Medical Education and Designated Institutional Official, Professor of Surgery, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-25-00212
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participant who underwent liver resection: Adult patients who underwent liver resection between January 2022 and December 2023. Data obtained from the American College of Surgeons National Surgical Quality Improvement Program (NSQIP)

SUMMARY:
A retrospective cohort study was conducted using the American College of Surgeons National Surgical Quality Improvement Program (NSQIP) database to identify adult patients who underwent liver resection between 2022 and 2023. Primary outcomes included 30-day mortality, sepsis, septic shock, readmission, and reoperation.

ELIGIBILITY:
Inclusion Criteria:

- Retrospective patients with condition only

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants wit hepatic neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 9411 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Number of deaths at 30 days
Number of participants with Sepsis | 30 days
  Number of participants with sepsis at 30 days
Number of participants with Septic Shock | 30 days
  Number of participants with septic shock at 30 days
Number of readmissions | 30 days
  Number of participants who had a remission at 30 days
Number of reoperations | 30 days
  Number of participants who had an reoperation at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leitman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Data are available indefinitely at (Link included in the URL field below).
URL: https://www.facs.org/quality-programs/data-and-registries/acs-nsqip/participant-use-data-file/